CLINICAL TRIAL: NCT01552525
Title: Regulation of L-Arginine Und Its Derivatives of Asymmetrical and Symmetrical Dimethylarginine and L-NG Monomethylarginine (ADMA/SDMA/L-NMMA) in Acute Kidney Injury and Correlation to Cardiac, Renal and Vascular Function and Mortality
Brief Title: L-Arginine, Symmetrical and Asymmetrical Dimethylarginine (SDMA/ADMA) in Acute Kidney Injury (AKI)
Status: Completed | Type: Observational
Sponsor: Wuerzburg University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 91/10
Record Dates: First submitted 2012-02-02; First posted 2012-03-13 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2012-03

CONDITIONS: Acute Kidney Injury
Keywords: acute kidney injury; asymmetric dimethylarginine; symmetric dimethylarginine; l-arginine; arterial stiffness; augmentation index; pulse wave velocity
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and urine samples will be centrifuged. One ml aliquots of plasma, serum, urine and a whole blood sample will be stored at -80°C.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- acute kidney injury: Patients with acute kidney injury according to the definition of AKIN (Acute Kidney Injury Network)

SUMMARY:
The purpose of the study is to determine the association between acute kidney injury and serum levels symmetrical and asymmetrical dimethylarginine (SDMA/ADMA) and their assumptive influence on mortality, renal function and on arterial stiffness.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) is a frequent complication with severe implications deteriorating overall prognosis. Nitric oxide (NO)-signal transduction plays an important role in mediating renal damage. NO is produced by NO-synthase (NOS) with L-arginine as its substrate. Endogenous L-Arginine derivatives, asymmetric and symmetric dimethylarginines (ADMA/SDMA), inhibit NO-production directly (AMDA) by blocking NOS activity or indirectly (SDMA) by blocking cellular L-Arginine uptake.

It is well known that SDMA and ADMA are markers of renal function (SDMA) and cardiovascular risk (ADMA/SDMA) in patients with chronic kidney disease (CKD). Moreover, ADMA and SDMA possibly even trigger cardiovascular risk in patients with CKD. However, there is only little information about the regulation and the influence of ADMA/SDMA in acute kidney injury.

ELIGIBILITY:
Inclusion Criteria:

* acute kidney injury according to the definition of AKIN (Acute Kidney Injury Network)
* no started renal replacement therapy (e.g. dialysis)

Exclusion Criteria:

* dialysis or continuous venovenous hemofiltration before recruitment
* no recovery from kidney injury according to the definition of AKIN (Acute Kidney Injury Network)
* palliative care
* life expectancy is severely limited (< six months) due to preexisting malignancy or other disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with acute kidney injury in the University Hospital of Wuerzburg will be recruited on the wards and in the emergency unit when nephrologists are consulted.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2011-01; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Difference in serum ADMA level between acute kidney injury and renal recovery | participants will be followed from the time of recruitment to the end of hospital stay, an expected average of 2 weeks
Difference in serum SDMA level between acute kidney injury and renal recovery | participants will be followed from the time of recruitment to the end of hospital stay, an expected average of 2 weeks

SECONDARY OUTCOMES:
Associations between ADMA/SDMA serum level and all cause mortality | participants will be followed from the time of recruitment to the end of hospital stay, an expected average of 2 weeks
Associations between ADMA/SDMA serum level and parameters of arterial stiffness | participants will be followed from the time of recruitment to the end of hospital stay, an expected average of 2 weeks
  Parameters of arterial stiffness include augmentation index and pulse wave velocity
Associations between ADMA/SDMA serum level and parameters of renal function | participants will be followed from the time of recruitment to the end of hospital stay, an expected average of 2 weeks
  Parameters of renal function include serum creatinine and estimated Glomerular Filtration Rate (eGFR)

CONTACTS AND LOCATIONS:
Overall Officials: Boris B Betz, Dr, Principal Investigator — Division of Nephrology Department of Medicine I University Hospital of Wuerzburg
Locations (1):
- University Hospital of Wuerzburg, Würzburg, Germany

REFERENCES:
- [Background] Mehta RL, Kellum JA, Shah SV, Molitoris BA, Ronco C, Warnock DG, Levin A; Acute Kidney Injury Network. Acute Kidney Injury Network: report of an initiative to improve outcomes in acute kidney injury. Crit Care. 2007;11(2):R31. doi: 10.1186/cc5713. PMID 17331245